CLINICAL TRIAL: NCT03593200
Title: Phase IIa, Open Label, Multiple Dose Study to Assess the Safety, Efficacy and Pharmacokinetics of Subcutaneously Administered APL-2 in Subjects With Paroxysmal Nocturnal Hemoglobinuria (PNH).
Brief Title: A Phase IIa Study to Assess the Safety, Efficacy, and Pharmacokinetics of Subcutaneously Administered Pegcetacoplan (APL-2) in Subjects With PNH
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Apellis Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: APL2-202
Record Dates: First submitted 2018-06-28; First posted 2018-07-20 (Actual); Results first posted 2020-12-22 (Actual); Last update posted 2020-12-22 (Actual); Status verified 2020-12

CONDITIONS: PNH
Keywords: PNH; Paroxysmal Nocturnal Hemoglobinuria; Complement inhibitor; Anemia; Hemoglobinuria; Hemolysis; Hematologic diseases; Extravascular hemolysis (EVH); Intravascular hemolysis (IVH); C3 inhibitor
MeSH Terms: conditions — Hemoglobinuria, Paroxysmal; Anemia; Hemoglobinuria; Hemolysis; Hematologic Diseases | interventions — pegcetacoplan

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Experimental: Cohort 1 (Experimental): 270 mg/day (up to 360 mg/day from Day 29) from Day 1 to Day 364*
  Interventions: Drug: Pegcetacoplan

INTERVENTIONS:
Drug: Pegcetacoplan — Complement (C3) Inhibitor
  Other Names: APL-2

SUMMARY:
This is a Phase IIa, open-label, multiple dose, study in patients with PNH who have not received eculizumab (Soliris ®) in the past. A single cohort of subjects is planned for evaluation.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years old (inclusive)
* Diagnosed with PNH (white blood cell (WBC) clone >10%)
* Lactose dehydrogenase (LD) ≥2 times the upper limit of normal
* Screening Ferritin ≥ normal and Total Iron Binding Capacity (TIBC) < LLN based on central lab reference ranges. If a subject is receiving iron supplements at screening, the investigator must ensure that his/her dose has been stable for 8 weeks prior to enrolment and must be maintained throughout the study
* Last transfusion within 12 months prior to screening
* Platelet count of >30,000/mm3 at the screening visit
* Absolute neutrophil count >500/ mm3 at the screening visit
* Women of child-bearing potential (WOCBP) must have a negative pregnancy test at screening and must agree to use protocol defined methods of contraception for the duration of the study
* Males must agree to use protocol defined methods of contraception and agree to refrain from donating sperm for the duration of the study
* Vaccination against Neisseria meningitides types A, C, W, Y and B, Streptococcus pneumoniae and Haemophilus influenzae Type B (Hib) either within 2 years prior to Day 1 dosing, or within 14 days after starting treatment with pegcetacoplan. Unless documented evidence exists that subjects are non-responders to vaccination as evidenced by titers or display titer levels within acceptable local limits
* Willing and able to give informed consent

Exclusion Criteria:

* Prior eculizumab (Soliris®) treatment
* Active bacterial infection
* Hereditary complement deficiency
* History of bone marrow transplantation
* Concurrent severe aplastic anemia (SAA), defined as currently receiving immunosuppressive therapy for SAA including but not limited to cyclosporin A, tacrolimus, mycophenolate mofetil or anti-thymocyte globulin
* Participation in any other investigational drug trial or exposure to another investigational agent, device or procedure within 30 days
* Evidence of QTcF prolongation defined as >450 ms for males and >470 ms for females at screening
* Breast-feeding women
* History of meningococcal disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2018-08-16 (Actual); Primary Completion 2019-10-22 (Actual); Study Completion 2019-10-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Federico Grossi, MD, PhD, Study Director — Study Director
Locations (3):
- Bulgaria (2):
  - Acibadem City Clinic MHAT Tokuda EAD Sofia, Sofia
  - Specialized Hospital for Active Treatment of Hematologic Diseases EAD, Sofia, Sofia
- Klinički centar Srbije, Belgrade, Serbia

REFERENCES:
- [Derived] Wong RSM, Pullon HWH, Amine I, Bogdanovic A, Deschatelets P, Francois CG, Ignatova K, Issaragrisil S, Niparuck P, Numbenjapon T, Roman E, Sathar J, Xu R, Al-Adhami M, Tan L, Tse E, Grossi FV. Inhibition of C3 with pegcetacoplan results in normalization of hemolysis markers in paroxysmal nocturnal hemoglobinuria. Ann Hematol. 2022 Sep;101(9):1971-1986. doi: 10.1007/s00277-022-04903-x. Epub 2022 Jul 22. PMID 35869170

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This Phase 2a, open-label, multiple-dose study was conducted in subjects with paroxysmal nocturnal hemoglobinuria (PNH) who had not received treatment with eculizumab (Soliris®) in the past, between 16 August 2018 and 22 October 2019.
Pre-assignment Details: Up to 20 subjects were planned to be enrolled; however, the sponsor decided to close recruitment after 4 subjects were enrolled based on the conclusion that sufficient data were collected to meet the study objectives.
Groups:
- Pegcetacoplan 270 mg/Day: Subjects received subcutaneous (SC) infusions of pegcetacoplan 270 milligrams (mg)/day up to Day 364. Intrasubject dose escalation up to a dosage of 360 mg/day was permitted if clinically indicated.
Period: Overall Study
Arm/Group | Pegcetacoplan 270 mg/Day
Started | 4
Completed (All subjects transitioned to an open-label extension study after Day 364.) | 4
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: The safety set consisted of all subjects who received at least 1 dose of study drug.
Groups:
- Pegcetacoplan 270 mg/Day: Subjects received SC infusions of pegcetacoplan 270 mg/day up to Day 364. Intrasubject dose escalation up to a dosage of 360 mg/day was permitted if clinically indicated.
Arm/Group | Pegcetacoplan 270 mg/Day
Number analyzed (Participants) | 4
Age, Continuous [Mean (Standard Deviation); unit: years] | 30.8 (11.81)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 1
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 4
  Not Hispanic or Latino | 4
Region of Enrollment [Number; unit: participants]
  Bulgaria | 2
  Serbia | 2

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects With Treatment Emergent Adverse Events (TEAEs) Including by Severity
Description: TEAEs were defined as adverse events (AE) that occurred after dosing on Day 1 and up to 30 days after the last dose of study drug. A treatment-related TEAE was defined as a TEAE with a relationship to study drug of possible, probable, or definite. TEAEs were graded according to the Common Terminology Criteria for Adverse Events (v4.03) based on: Grade 1: Mild, Grade 2: Moderate, Grade 3: Severe, Grade 4: Life-threatening, Grade 5: Death related to AE.
Time Frame: From Day 1 to 30 days after the last dose (approximately 56 weeks)
Population: The safety set consisted of all subjects who received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Pegcetacoplan 270 mg/Day
Number analyzed (Participants) | 4
Participants
  All TEAEs | 3
  Treatment-related TEAEs | 2
  Serious TEAEs | 1
  TEAEs leading to study drug discontinuation | 0
  TEAEs with mild intensity | 2
  TEAEs with moderate intensity | 0
  TEAEs with severe intensity | 1
  TEAEs with life threatening intensity | 0
  TEAEs leading to death | 0

2. Primary Outcome: Mean Change From Baseline in Lactate Dehydrogenase (LDH) Level
Description: Serum chemistry assessments of LDH were made at the last measurement prior to the first dose of pegcetacoplan (baseline) and periodically throughout the treatment period.
Time Frame: Baseline and Day 365
Population: The Intent-to-treat (ITT) set consisted of all subjects who received at least 1 dose of study drug.
Measure: Mean (Standard Deviation); unit: units/liter
Arm/Group | Pegcetacoplan 270 mg/Day
Number analyzed (Participants) | 4
units/liter | -2322.8 (635.41)

3. Primary Outcome: Mean Change From Baseline in Haptoglobin Level
Description: Serum chemistry assessments of haptoglobin were made at the last measurement prior to the first dose of pegcetacoplan (baseline) and periodically throughout the treatment period.
Time Frame: Baseline and Day 365
Population: The ITT set consisted of all subjects who received at least 1 dose of study drug.
Measure: Mean (Standard Deviation); unit: grams/liter
Arm/Group | Pegcetacoplan 270 mg/Day
Number analyzed (Participants) | 4
grams/liter | 0.08 (0.150)

4. Primary Outcome: Mean Change From Baseline in Hemoglobin (Hb) Level
Description: Hematology assessments of Hb were made at the last measurement prior to the first dose of pegcetacoplan (baseline) and periodically throughout the treatment period.
Time Frame: Baseline and Day 365
Population: The ITT set consisted of all subjects who received at least 1 dose of study drug.
Measure: Mean (Standard Deviation); unit: grams/deciliter
Arm/Group | Pegcetacoplan 270 mg/Day
Number analyzed (Participants) | 4
grams/deciliter | 5.27 (1.875)

5. Secondary Outcome: Mean Change From Baseline in Functional Assessment of Chronic Illness Therapy (FACIT)-Fatigue Score
Description: The FACIT-Fatigue scale is a 13 item Likert scaled instrument where the subject was presented with 13 statements and asked to indicate their response as it applied to the past 7 days. The 5 possible responses were 'Not at all' (0), 'A little bit (1), 'Somewhat' (2), 'Quite a bit' (3) and 'Very much' (4). With 13 statements the total score had a range of 0 to 52. Higher score corresponds to a higher quality of life (QoL).
Time Frame: Baseline and Day 365
Population: The ITT set consisted of all subjects who received at least 1 dose of study drug.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Pegcetacoplan 270 mg/Day
Number analyzed (Participants) | 4
score on a scale | 6.5 (5.45)

6. Secondary Outcome: Mean Change From Baseline in Absolute Reticulocyte Count (ARC) Level
Description: Hematology assessments of ARC were made at the last measurement prior to the first dose of pegcetacoplan (baseline) and periodically throughout the treatment period.
Time Frame: Baseline and Day 365
Population: The ITT set consisted of all subjects who received at least 1 dose of study drug.
Measure: Mean (Standard Deviation); unit: ARC/nanoliter
Arm/Group | Pegcetacoplan 270 mg/Day
Number analyzed (Participants) | 4
ARC/nanoliter | -144.3 (98.51)

7. Secondary Outcome: Mean Change From Baseline in Total Bilirubin Level
Description: Serum chemistry assessments of total bilirubin were made at the last measurement prior to the first dose of pegcetacoplan (baseline) and periodically throughout the treatment period.
Time Frame: Baseline and Day 365
Population: The ITT set consisted of all subjects who received at least 1 dose of study drug.
Measure: Mean (Standard Deviation); unit: micromoles/liter
Arm/Group | Pegcetacoplan 270 mg/Day
Number analyzed (Participants) | 4
micromoles/liter | -21.53 (8.358)

8. Secondary Outcome: Mean Number of Red Blood Cell (RBC) Transfusions Per Month
Description: The number of on-study RBC transfusions was monitored throughout the treatment period.
Time Frame: From Day 1 to Day 364
Population: The ITT set consisted of all subjects who received at least 1 dose of study drug.
Measure: Mean (Full Range); unit: transfusions
Arm/Group | Pegcetacoplan 270 mg/Day
Number analyzed (Participants) | 4
transfusions | 0 [0 to 0]

9. Secondary Outcome: Mean Change From Baseline in Linear Analog Scale Assessment (LASA) Score for QoL
Description: The LASA consists of 3 items, where the respondents were asked to rate their perceived level of functioning. Specific domains included activity level, ability to carry out daily activities, and an item for overall QoL. Their level of functioning was reported on a 0 to 100 scale with 0 indicates "As low as could be" and 100 indicates "As high as could be". The combined score ranged from 0 to 300, with higher scores corresponding to a higher QoL.
Time Frame: Baseline and Day 365
Population: The ITT set consisted of all subjects who received at least 1 dose of study drug.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Pegcetacoplan 270 mg/Day
Number analyzed (Participants) | 4
score on a scale | 66.5 (55.75)

10. Secondary Outcome: Mean Serum Concentrations of Pegcetacoplan
Description: Serum concentrations of pegcetacoplan at Day 365 are presented.
Time Frame: Day 365
Population: The Pharmacokinetic (PK) set consisted of all subjects in the safety set who had at least 1 quantifiable PK sample post dose PK measurement.
Measure: Mean (Standard Deviation); unit: microgram per milliliter (ug/mL)
Arm/Group | Pegcetacoplan 270 mg/Day
Number analyzed (Participants) | 4
microgram per milliliter (ug/mL) | 622.0 (92.13)

11. Secondary Outcome: Mean Area Under the Serum Concentration Versus Time Curve From Time 0 to the Last Measurable Concentration at the End of the Study (AUCtotal)
Description: The AUCtotal of pegcetacoplan was estimated using a non-compartmental approach.
Time Frame: Blood samples were collected predose and at least 2.5 hours post dose on Day 1 and predose on Days 2 up to Day 365.
Population: The PK set consisted of all subjects in the safety set who had at least 1 quantifiable PK sample post dose PK measurement.
Measure: Mean (Standard Deviation); unit: hour*ug/mL
Arm/Group | Pegcetacoplan 270 mg/Day
Number analyzed (Participants) | 4
hour*ug/mL | 5818803.2534 (975444.77662)

12. Secondary Outcome: Mean Maximum Observed Predose Serum Concentration During the Study (Ctrough,Max,Total)
Description: The Ctrough,max,total of pegcetacoplan was estimated using a non-compartmental approach.
Time Frame: Blood samples were collected predose and at least 2.5 hours post dose on Day 1 and predose on Days 2 up to Day 365.
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: ug/mL
Arm/Group | Pegcetacoplan 270 mg/Day
Number analyzed (Participants) | 4
ug/mL | 783.5 (116.25)

ADVERSE EVENTS:
Time Frame: TEAEs were collected from Day 1 up to 30 days after the last dose of study drug (a total of approximately 56 weeks).
Description: The safety set consisted of all subjects who received at least 1 dose of study drug.
Arm/Group | Pegcetacoplan 270 mg/Day
All-Cause Mortality (participants affected / at risk) | 0/4
Serious Adverse Events (participants affected / at risk) | 1/4
Other Adverse Events (participants affected / at risk) | 3/4
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pegcetacoplan 270 mg/Day (N=4)
Rib fracture (Injury, poisoning and procedural complications) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pegcetacoplan 270 mg/Day (N=4)
Administration site swelling (General disorders) | 1 (1)
Injection site discolouration (General disorders) | 1 (1)
Injection site erythema (General disorders) | 1 (8)
Injection site pruritus (General disorders) | 1 (1)
Injection site swelling (General disorders) | 1 (4)
Dizziness (Nervous system disorders) | 2 (3)
Erythema (Skin and subcutaneous tissue disorders) | 2 (37)
Rhinitis (Infections and infestations) | 1 (2)
Scrotal irritation (Reproductive system and breast disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
Given the small sample size, no conclusions should be drawn from the results summarized and reported as descriptive statistics in Outcome Measures 9-12.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2018-01-31): https://cdn.clinicaltrials.gov/large-docs/00/NCT03593200/Prot_000.pdf
  • Statistical Analysis Plan (2019-07-17): https://cdn.clinicaltrials.gov/large-docs/00/NCT03593200/SAP_001.pdf